CLINICAL TRIAL: NCT05972980
Title: Ventilator-Associated Pneumonia and Multidrug-Resistant Pathogens: A Prospective Observational Monocentric Comparative Study Between Critically Ill Non-COVID-19 and COVID-19 Patients
Brief Title: Ventilator-Associated Pneumonia in Critically Ill COVID-19 vs. Non-COVID-19 Patients
Status: Completed | Type: Observational
Sponsor: University of Turin, Italy (Other)
Responsible Party: Sponsor
Other Study IDs: MR-VAP-C19
Record Dates: First submitted 2023-07-31; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Infections; Critical Illness; Superinfection; Organ Failure, Multiple; Ventilator Associated Pneumonia; Septic Shock
MeSH Terms: conditions — Infections; Critical Illness; Superinfection; Multiple Organ Failure; Pneumonia, Ventilator-Associated; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-COVID-19 cohort: Patients with Ventilator Acquired Pneumonia without COVID-19.
  The patients belonging to the NON-COVID cohort were admitted to three intensive care units at Molinette Hospital (Turin, Italy):
  * General Intensive Care Unit - admitting primarily medically critical patients and a smaller proportion of surgical patients, originating from the Hospital's Emergency Department or other Intensive Care Units in Piedmont. It serves as the regional referral center for Extracorporeal Membrane Oxygenation (ECMO).
  * Emergency Department - Intensive Care Unit (PSAR) - admitting both medical and surgical patients in urgent conditions.
  * Cardiac - Intensive Care Unit- admitting patients undergoing elective or emergency cardio-surgical interventions, and serving as a referral center for heart and lung transplants and the implantation of external ventricular assists.
- COVID-19 cohort: Patients with Ventilator Acquired Pneumonia with COVID-19. Confirmation of pneumonia was achieved by using the Reverse Transcriptase-Polymerase Chain Reaction (RT-PCR) technique on a sample collected from the lower respiratory tract.
  The COVID-19 cohort consists of patients admitted at the "Città della Salute e della Scienza" University Hospital (Turin, Italy) in two intensive care units at Molinette Hospital, dedicated to treating critically ill patients with COVID-19.
  Interventions: Other: COVID-19

INTERVENTIONS:
Other: COVID-19 — The investigators stratified our population based on COVID-19 virus positivity to identify any risk factors in this population compared to the NON-COVID-19 population.
  Groups: COVID-19 cohort

SUMMARY:
The COVID-19 pandemic has led to an increased incidence of ventilator-associated pneumonia (VAP) among critically ill patients. However, in a context of high prevalence of multidrug-resistant organisms (MDROs) there is a lack of direct comparison between the incidence of VAP in COVID-19 and non-COVID-19 cohorts.

The investigators conducted a prospective, single-center cohort study comparing COVID-19 patients admitted to the intensive care unit (ICU) of the Città della Salute e della Scienza University Hospital in Turin, Italy, between March 2020 and December 2021 (COVID-19 group), with a historical cohort of ICU-mixed patients admitted between June 2016 and March 2018 (NON-COVID-19 group).

DETAILED DESCRIPTION:
The study aims to explore the occurrence and characteristics of ventilator-associated pneumonia (VAP) in critically ill patients during two distinct periods: the pre-pandemic era and the COVID-19 pandemic. VAP, a serious complication arising from invasive mechanical ventilation (IMV) lasting at least 48 hours, had a crude incidence of 5% to 40% before the COVID-19 pandemic, whereas COVID-19 patients experienced even higher rates, reaching 48-64%.

The COVID-19 pandemic triggered an unprecedented rise in ICU admissions due to severe acute respiratory syndrome caused by the SARS-CoV-2 virus, leading to a considerable number of patients requiring IMV. Mechanical ventilation is a known risk factor for VAP, and COVID-19 exacerbates this risk due to factors like disease-induced immunoparalysis, prolonged mechanical ventilation and sedation, and more frequent application of prone positioning.

Despite the widespread need for prolonged mechanical ventilation in COVID-19 patients, few studies have compared the impact of VAP between pre-pandemic and COVID-19 populations. Additionally, limited research exists on the risk factors for VAP development in COVID-19 patients and the use of scoring systems like SAPS and SOFA as prognostic factors in this specific context. Although the coVAPid study offered insights into VAP risk factors in COVID-19 patients compared to those with influenza, it inadequately addressed the prevalence of multidrug-resistant organisms (MDROs) in this population, particularly carbapenem-resistant Acinetobacter baumannii (CR-Ab). Hence, this study aims to bridge this knowledge gap by investigating VAP's impact in a setting characterized by a high incidence of multidrug resistance.

To achieve this, the study will take place at the Molinette Hospital of the "Città della Salute e della Scienza" University Hospital in Turin, Italy, over a six-year period, spanning from January 2016 to December 2022. This retrospective, observational, and monocentric study will focus on two distinct cohorts: the pre-pandemic cohort (NON-COVID-19) and the COVID-19 cohort.

Researchers will identify ventilator-associated pneumonia (VAP) episodes based on the current definitions provided by the European Center for Disease Prevention and Control (ECDC). Patients will be monitored until hospital discharge to assess outcomes, including ICU mortality, overall mortality, duration of ICU stay, and duration of hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients diagnosed with ventilator-associated pneumonia
* Patients admitted to the intensive care units
* Patients who underwent mechanical ventilation for a duration longer than 48 hours

Exclusion Criteria:

* Patients in extreme end-of-life conditions
* Pregnant individuals
* Patients under 18 years of age
* Patients who did not meet the diagnosis criteria for ventilator-associated pneumonia
* Patients who underwent mechanical ventilation for a duration equal to or shorter than 48 hours
* Ventilator-associated tracheobronchitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients diagnosed with ventilator-acquired pneumonia admitted to the intensive care unit of the primary hospital "Molinette," Città della Salute e della Scienza, Turin, Italy.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-01-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Mortality | 28 days
  Mortality within the first 28 days from ICU admission

SECONDARY OUTCOMES:
ICU mortality | From date of enrollment until the date of intensive care unit discharge, assessed up to 6 months
  Mortality during intensive care unit stay
Hospital mortality | From date of enrollment until the date of hospital discharge, assessed up to 6 months
  Mortality during hospital stay
Mechanical ventilation days | From date of enrollment until the date of intensive care unit discharge, assessed up to 6 months
  Days of mechanical ventilation length of stay
Ventilator acquired pneumonia incidence | From date of enrollment until the date of intensive care unit discharge, assessed up to 6 months
  Incidence of ventilator acquired pneumonia
Ventilator acquired pneumonia incidence | 28 days
  Incidence of ventilator acquired pneumonia
Multidrug-resistant micro-organisms incidence | From date of enrollment until the date of intensive care unit discharge, assessed up to 6 months
  Incidence of Multidrug-resistant micro-organisms
Difficult to treat pathogens incidence | From date of enrollment until the date of intensive care unit discharge, assessed up to 6 months
  Incidence of difficult to treat pathogens
Hospital length of stay | From date of enrollment until the date of hospital discharge, assessed up to 6 months
  Duration of hospital length of stay
Intensive care unit length of stay | From date of enrollment until the date of intensive care unit discharge, assessed up to 6 months
  Duration of intensive care unit length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Luca Brazzi, Study Chair — University of Torino
Locations (1):
- AOU Città della Salute e della Scienza di Torino, Torino, Italy